CLINICAL TRIAL: NCT02508168
Title: An Open-Label, Single-dose, Randomized, Crossover Study to Determine the Bioavailability and Bioequivalence of Alogliptin 12.5 mg and Metformin 1000 mg When Administered as Individual Tablets and as a Fixed-Dose Combination Tablet Vipdomet (Alogliptin FDC With Metformin) in Russian Healthy Subjects
Brief Title: Phase 1 Bioavailability Study of SYR-322MET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SYR-322MET-1003; U1111-1168-6473 (Registry Identifier: WHO)
Record Dates: First submitted 2015-07-23; First posted 2015-07-24 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy
MeSH Terms: interventions — alogliptin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence I: AB (Experimental): SYR-322MET (alogliptin 12.5 mg and metformin 1000 mg) fixed-dose combination (FDC) tablets, orally, once, on Day 1 of Period 1, followed by a 7-day washout period, followed by alogliptin 12.5 mg tablets and metformin 1000 mg tablets, orally, once, on Day 1 of Period 2.
  Interventions: Drug: Alogliptin; Drug: Metformin Hydrochloride; Drug: SYR-322MET
- Sequence II: BA (Experimental): Alogliptin 12.5 mg tablets, orally and metformin 1000 mg tablets, orally, once, on Day 1 of Period 1, followed by a 7-day washout period, followed by SYR-322MET (alogliptin 12.5 mg and metformin 1000 mg) fixed-dose combination (FDC) tablets, orally, once, on Day 1 of Period 2.
  Interventions: Drug: Alogliptin; Drug: Metformin Hydrochloride; Drug: SYR-322MET

INTERVENTIONS:
Drug: Alogliptin — Alogliptin 12.5 mg tablets
  Other Names: Vipidia
Drug: Metformin Hydrochloride — Metformin hydrochloride 1000 mg tablets
  Other Names: Glucophage
Drug: SYR-322MET — SYR-322MET (alogliptin 12.5 mg and metformin 1000 mg) fixed-dose combination (FDC) tablets

SUMMARY:
The purpose of this study is to determine the relative bioavailability of alogliptin 12.5 milligram (mg) and immediate-release metformin 1000 mg when administered as individual tablets and as a fixed-dose combination (FDC) product.

DETAILED DESCRIPTION:
The drug being tested in this study is called SYR-322MET (alogliptin 12.5 mg and metformin 1000 mg FDC tablet). SYR-322MET is being tested to assess whether its pharmacokinetic properties (how it is processed by the body) are affected when administered as a FDC compared to administration of alogliptin and metformin alone. This study will look at lab results in people who take SYR-322MET.

This crossover study will enroll approximately 24 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of two treatment sequences. All participants will receive both treatments over two periods; the order of receipt will be determined by the randomization code. All participants will receive the following study medications by the end of the study:

* Alogliptin 12.5 mg + Metformin 1000 mg as individual tablets
* SYR-322MET (alogliptin 12.5 mg and metformin 1000 mg fixed-dose combination [FDC] tablet)

This single center trial will be conducted in Russia. The overall time to participate in this study is up to 63 days. Participants will make multiple visits to the clinic including two 4-day periods of confinement to the clinic, and will be contacted by telephone 14 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. Signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures including requesting that a participant fast for any laboratory evaluations.
3. Is a healthy male or female.
4. Is aged 18 to 55 years, inclusive, at the time of informed consent and first study medication dose.
5. Weighs at least 50 kilogram (kg) and has a body mass index (BMI) from 18.5 to 30.0 kilogram per square meter (kg/m^2), inclusive at Screening.
6. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 30 days after last dose.
7. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent and throughout the duration of the study and for 30 days after last dose.

Exclusion Criteria

1. Has received any investigational compound within 30 days prior to Check-in (Day-1).
2. Has received alogliptin or metformin hydrochloride (HCl) in a previous clinical study or as a therapeutic agent within 90 days prior to Check-in (Day-1).
3. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (example, spouse, parent, child, sibling) or may consent under duress.
4. Has clinically significant history or current diagnosis of cardiovascular, respiratory, neurological, endocrine, hematopoietic, immune, urinary, genital, gastrointestinal, hepatic and psychiatric diseases.
5. Has fasting blood glucose lower than 3.88 millimoles per liter (mmol/L)
6. Has experienced acute infectious diseases within 4 weeks before screening.
7. Has a history of clinically significant allergic reactions or has a known hypersensitivity to any component of the formulation of alogliptin, metformin or related compounds.
8. Has a positive urine drug result for drugs of abuse (defined as any illicit drug use) or positive alcohol breath test at Screening or Check-in (Day -1).
9. Consumes over 10 drinks weekly (1 drink is equivalent to 0.5 liters of beer, 200 milliliter [mL] of dry wine or 50 mL of hard liquor) or has a history of alcoholism, drug and/or substance abuse.
10. Has taken any excluded medication, supplements, or food products during the time periods listed in the Excluded Medications and Dietary Products table, including intake of medicines with pronounced effects on blood circulation, liver function (barbiturates, omeprazole, cimetidine, etc.) within 2 months before Day -1 of Period 1.
11. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 30 days after participating in this study; or intending to donate ova during such time period.
12. If male, the participant intends to donate sperm during the course of this study or for 12 weeks after the last dose of study medication.
13. If female, the subject is having unprotected sex with non-sterilized men within 30 days before the IMP administration.
14. Has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (that is, a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis, frequent [more than once per week] occurrence of heartburn, or any surgical intervention.
15. Has non-standard diet (example, vegetarian or vegan) or lifestyle (including nighttime work, extreme physical activity such as weights lifting), which may interfere with the trial.
16. Has a history of cancer, except basal cell carcinoma which has been in remission for at least 5 years prior to Day 1 of Period 1.
17. Has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody or syphilis at screening.
18. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to Check-in Day -1. Cotinine test is positive at Screening or Check-in (Day 1).
19. Has poor peripheral venous access.
20. Has donated or lost 450 mL or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 30 days prior to Day 1 of Period 1.
21. Has abnormalities in routine physician examination, laboratory and/or ECG findings
22. Has a systolic blood pressure greater (>)130 millimeter of mercury (mm Hg) or less than (<)100 mm Hg , diastolic blood pressure >90 mm Hg or <70 mm Hg; heart rate <60 bpm or >80 bpm at screening (Day -28 to Day -2) or check-in to Period 1 (Day -1).
23. Has participated in any clinical study within 3 months before Day -1 of Period 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
AUC(0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Alogliptin | Day 1 predose and at multiple time points (up to 72 hours) post-dose.
  (AUC(0-tlqc) is a measure of total plasma exposure to the drug from Time 0 to Time of the Last Quantifiable Concentration (AUC[0-tlqc]).
Cmax: Maximum Observed Plasma Concentration for Alogliptin | Day 1 predose and at multiple time points (up to 72 hours) post-dose.
  Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
AUC(0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Metformin | Day 1 predose and at multiple time points (up to 72 hours) post-dose.
  (AUC(0-tlqc) is a measure of total plasma exposure to the drug from Time 0 to Time of the Last Quantifiable Concentration (AUC[0-tlqc]).
Cmax: Maximum Observed Plasma Concentration for Metformin | Day 1 predose and at multiple time points (up to 72 hours) post-dose.
  Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.

SECONDARY OUTCOMES:
Percentage of Participants who Experience at Least one Post-dose Adverse Event (AE) | Day 1 of Period 1 up to 30 days after the last dose of study medication (up to 38 days)
  An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug.
Percentage of Participants who Meet the Markedly Abnormal Criteria for Safety Laboratory Tests at Least Once Post Dose | At Day 4 and Day 7 of Period 2
  Standard safety laboratory values (hematology and chemistry) will be collected throughout study and compared to pre-specified criteria for markedly abnormal values.
Percentage Of Participants who Meet the Markedly Abnormal Criteria for Vital Sign Measurements at Least Once Post Dose | Day 1 up to Day 4 of each period
  Vital sign measurements will be collected throughout study and compared to pre-specified criteria for markedly abnormal values.
Percentage of Participants who Meet the Markedly Abnormal Criteria for Safety Electrocardiogram (ECG) Parameters at Least Once Post Dose | At Day 1 and Day 4 of each period
  Standard 12-lead ECG measurements will be collected throughout the study and compared to pre-specified criteria for markedly abnormal values.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda